CLINICAL TRIAL: NCT00658996
Title: A Study to Evaluate the Product Performance of a Prism-Ballasted Toric Contact Lens When Worn by Currently Adapted Soft Contact Lens Wearers.
Brief Title: Product Performance of a Toric Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 559
Record Dates: First submitted 2008-04-12; First posted 2008-04-16 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SofLens DD Toric (Experimental): Bausch & Lomb SofLens Daily Disposable Toric Contact Lens
  Interventions: Device: SofLens DD Toric
- Ciba Vision Toric Lens (Active Comparator): Ciba Vision Focus Dailies Toric Contact Lens
  Interventions: Device: Ciba Vision Focus Dailies Toric Contact Lens

INTERVENTIONS:
Device: SofLens DD Toric — daily disposable wear contact lens for 2 weeks
  Arms: SofLens DD Toric
Device: Ciba Vision Focus Dailies Toric Contact Lens — daily disposable wear contact lens for 2 weeks
  Arms: Ciba Vision Toric Lens

SUMMARY:
Product performance of a Bausch & Lomb Toric Contact Lens compared to Ciba Vision Focus Daily Toric Contact Lens

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adapted soft contact lens wearer with astigmatism of 0.50 Diopter or greater
* Visual acuity (VA) correctable to 0.3 logMar or better (driving vision)
* Clear central cornea

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using systemic or topical medications
* Wears monovision or multifocal contact lenses
* Any grade 2 or greater slit lamp findings
* Adapted wearer of Ciba Focus Dailies Toric lens upon study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, PhD,MCOptom, Study Director — Bausch & Lomb Incorporated; Benny Chian, MCOptom,DO, Principal Investigator — Laser Focus Sdn Bhd, Vision Correction Centre
Locations (1):
- Laser Focus Sdn Bhd, Vision Correction Centre, Johor Bahru, Malaysia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 4-week study was conducted at 12 sites in Asia. First participant enrolled 4/16/08, last participant visit was 6/20/08
Pre-assignment Details: 220 participants were enrolled in the study, 4 participants were ineligible at screening visit, 216 Subjects started the first intervention. 211 participants started the second intervention. 209 participants completed the study.
Groups:
- SofLens DD Toric First, Then Focus Dailies Toric: Bausch & Lomb SofLens Daily Disposable Toric Contact Lens first then crossover to Ciba Vision Focus Dailies Toric Lens
- Focus Dailies Toric First, Then SofLens DD Toric: Ciba Vision Focus Dailies Toric Lens first, then crossover to Bausch & Lomb SofLens Daily Disposable Toric Contact Lens
Period: First Intervention
Arm/Group | SofLens DD Toric First, Then Focus Dailies Toric | Focus Dailies Toric First, Then SofLens DD Toric
Started | 109 | 107
Completed | 108 | 106
Not Completed | 1 | 1
Not completed — Positive slit lamp finding | 1 | 0
Not completed — Lack of lenses | 0 | 1
Period: Crossover Period
Arm/Group | SofLens DD Toric First, Then Focus Dailies Toric | Focus Dailies Toric First, Then SofLens DD Toric
Started | 108 | 106
Completed | 106 | 105
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Ineligible | 1 | 1
Period: Second Intervention
Arm/Group | SofLens DD Toric First, Then Focus Dailies Toric | Focus Dailies Toric First, Then SofLens DD Toric
Started | 106 | 105
Completed | 105 | 104
Not Completed | 1 | 1
Not completed — Developed a stye on upper lid | 1 | 0
Not completed — Positive slit lamp finding | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Population enrolled at start of study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 216
Age Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 216
  White | 0
  Black | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Symptoms and Complaints
Description: 1-100 Scale for each eye. Zero represented the least favorable rating and 100 represented the most favorable.
Time Frame: Over-all follow-up visits for 2 week period
Population: All eligible, dispensed eyes, Overall follow-up visits.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Units Other Than Participants: eyes
Groups:
- Focus Dailies Toric: Ciba Vision Focus Dailies Toric contact lenses
Arm/Group | SofLens DD Toric | Focus Dailies Toric
Number analyzed (Participants) | 213 | 210
Number analyzed (eyes) | 426 | 420
Scores on a Scale
  Comfort | 79.3 (17.1) | 77.7 (17.6)
  End of Day Comfort | 73.5 (19.6) | 71.5 (19.9)
  Lens Awareness | 78.8 (17.9) | 75.6 (20.4)
  Lens Cleanliness | 87.5 (12.7) | 86.5 (13.0)
  Irritation | 83.0 (15.6) | 79.3 (19.6)
  Itching | 86.4 (14.9) | 83.9 (17.2)
  Dryness | 77.4 (18.0) | 73.7 (20.3)
  Redness | 86.3 (14.9) | 81.5 (19.5)
  Vision | 77.1 (19.1) | 84.3 (14.6)
  Lens Handling | 87.4 (13.0) | 76.1 (21.2)
  Overall Impression | 78.7 (16.2) | 75.9 (17.5)

2. Secondary Outcome: Slit Lamp Findings
Description: Graded 0-4 where 0=none and 4=severe on measure of epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, superior tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates
Time Frame: Over-all follow-up visits, 2 weeks
Population: All dispensed eyes, over all follow-up visits
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | SofLens DD Toric | Focus Dailies Toric
Number analyzed (Participants) | 215 | 215
Number analyzed (eyes) | 430 | 430
Eyes
  Slit Lamp Findings > Grade 2 | 0 | 2
  Slit Lamp Findings </= Grade 2 | 430 | 428

3. Primary Outcome: Contact Lens High Contrast Visual Acuity
Description: VA measures at each scheduled visit were averaged to obtain an overall measure for each eye. A non-inferiority upper bound of 0.06 (3 letters) were used to assess the difference (Test - Control) in overall logMAR VA.
Time Frame: Over-all follow-up visits, 2 weeks
Population: All eligible, dispensed eyes
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | SofLens DD Toric | Focus Dailies Toric
Number analyzed (Participants) | 213 | 210
Number analyzed (eyes) | 426 | 420
LogMAR | -0.007 (0.0669) | -0.014 (0.0696)

ADVERSE EVENTS:
Time Frame: One month
Groups:
- Ciba Vision Toric Lens: Ciba Vision Focus Dailies Toric Lens
Arm/Group | SofLens DD Toric | Ciba Vision Toric Lens
Serious Adverse Events (participants affected / at risk) | 0/215 | 0/216
Other Adverse Events (participants affected / at risk) | 0/215 | 0/216

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other